CLINICAL TRIAL: NCT00772499
Title: Vascular Improvement With Olmesartan Medoxomil Study
Acronym: VIOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Director Medical Research, Daiichi Sankyo, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 866-432
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Olmesartan Medoxomil; Hydrochlorothiazide; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): olmesartan medoxomil tablets with added doses of hydrochlorothiazide, amlodipine, or hydralazine, if required to maintain target blood pressure
  Interventions: Drug: olmesartan medoxomil + hydrochlorothiazide + amlodipine + hydralazine if necessary to control blood pressure
- 2 (Active Comparator): Atenolol tablets with added doses of hydrochlorothiazide, amlodipine, or hydralazine, if required to maintain target blood pressure
  Interventions: Drug: atenolol+ hydrochlorothiazide + amlodipine + hydralazine if necessary to control blood pressure

INTERVENTIONS:
Drug: olmesartan medoxomil + hydrochlorothiazide + amlodipine + hydralazine if necessary to control blood pressure — Tablets and capsules for oral administration once or twice daily for up to 52 weeks
  Arms: 1
Drug: atenolol+ hydrochlorothiazide + amlodipine + hydralazine if necessary to control blood pressure — Tablets and capsules for oral administration once or twice daily for up to 52 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to compare in patients with primary hypertension, the non-blood pressure lowering effects of one-year therapy with olmesartan medoxomil vs. those of atenolol on changes in the vascular structure and function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18-75 years of age
* Mean seated diastolic BP 90-109 or mean seated systolic BP of 140-179

Exclusion Criteria:

* Secondary hypertension
* Renal disease
* Diabetes mellitus
* Serum creatinine >3.0 mg/dL
* Hemoglobin <10 mg/dL (males) or <9mg/dL (females)
* WBC count <2000 cells/mL
* Platelet count <100,000 cells/mL
* Either ALT & AST >2.5 x upper limit of normal
* BMI >35 kg/m2
* TIA or cerebrovascular attack within 3 months of study entry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2002-11; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Subcutaneous gluteal fat arteriole measurements prior to and after 52 weeks of therapy | 52 weeks

SECONDARY OUTCOMES:
Results of vascular function tests | 12 weeks
Results of vascular function tests | 28 weeks
Results of vascular function tests | 52 weeks
Measurement of serum lipid and markers of atherosclerosis | 12 weeks
Measurement of serum lipid and markers of atherosclerosis | 28 weeks
Measurement of serum lipid and markers of atherosclerosis | 52 weeks
Retinal arteriole measurements | 52 weeks
Calculation of insulin sensitivity measurement | 12 Weeks
Calculation of insulin sensitivity measurement | 28 weeks
Calculation of insulin sensitivity measurement | 52 weeks
24 hour urine creatinine and thromboxane B2 measurements | 12 weeks
Calculation of albumin-to-creatinine ratio and sodium-to-creatinine ratio | 12 weeks
Calculation of albumin-to-creatinine ratio and sodium-to-creatinine ratio | 28 weeks
Calculation of albumin-to-creatinine ratio and sodium-to-creatinine ratio | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina, United States